CLINICAL TRIAL: NCT06525246
Title: ONO-7475-03: ONO-7475 Phase I Study An Open-label, Uncontrolled Study of ONO-7475 in Combination With Osimertinib in EGFR Gene Mutation-positive Non-small Cell Lung Cancer
Brief Title: Study of ONO-7475 in Combination With Osimertinib in EGFR Gene Mutation-positive Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONO-7475-03; jRCT2051210045 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Stage IIIB Non-small Cell Lung Cancer; Stage IIIC Non-Small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer; Recurrent Non-Small Cell Lung Cancer; EGFR Mutation-Related Tumors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ONO-7475+Osimertinib (Experimental)
  Interventions: Drug: ONO-7475; Drug: Osimertinib Mesylate

INTERVENTIONS:
Drug: ONO-7475 — Specified dose, once daily
Drug: Osimertinib Mesylate — Specified dose, once daily

SUMMARY:
This study is to evaluate the tolerability and safety of ONO-7475 in combination with osimertinib in the first-line treatment of patients with EGFR-mutated, stage IIIB/IIIC/IV or recurrent non-small cell lung cancer (NSCLC), which is unsuitable for radical irradiation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stage IIIB/IIIC/IV or recurrent NSCLC, which is unsuitable for radical irradiation
2. Patients with confirmed EGFR gene exon 19 deletion or EGFR gene exon 21 mutation(L858R)and who are scheduled to receive osimertinib
3. Patient has an ECOG performance status of 0-1

Exclusion Criteria:

1. Patients with severe complication
2. Patients with multiple primary cancers

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities（DLT） Dose-limiting toxicities（DLT） Dose-limiting toxicities（DLT） | 28 days
Adverse event (AE) | Up to 28 days after the last dose

SECONDARY OUTCOMES:
Pharmacokinetics (Cmax) | Up to 57 Days
Pharmacokinetics (Tmax) | Up to 57 Days
Pharmacokinetics (AUC) | Up to 57 Days
Pharmacokinetics (Ctrough) | Up to 57 Days
Objective Response Rate (ORR) | Through study completion, an average of 2 year
Disease Control Rate (DCR) | Through study completion, an average of 2 year
Overall Survival (OS) | Through study completion, an average of 3 year
Progression-Free Survival (PFS) | Through study completion, an average of 2 year
Duration of Response (DOR) | Through study completion, an average of 2 year
Time to Response (TTR) | Through study completion, an average of 2 year
Best Overall Response (BOR) | Through study completion, an average of 2 year
Percent change in the sum diameters of the target lesions | Through study completion, an average of 2 year
Maximum percent change in the sum diameters of the target lesions | Through study completion, an average of 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (13):
- Japan (13):
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Hyogo College Of Medicine College Hospital, Nishinomiya, Hyōgo
  - Kitasato University Hospital, Sagamihara-shi, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Saitama Cancer Center, Ina, Kitaadati-gun, Saitama
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto, Kyoto
  - Osaka International Cancer Institute, Osaka, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki, Osaka
  - Shizuoka Cancer Center, Nagaizumi-chō, Sunto-gun, Shizuoka
  - The Cancer Institute Hospital Of JFCR, Koto-Ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-Ku, Tokyo
  - Nigata Cancer Center Hospital, Niigata

IPD SHARING:
Plan to Share IPD: No